CLINICAL TRIAL: NCT02192684
Title: Interfacing Adiposity, Sleep Apnea, and Insulin Resistance
Brief Title: Obesity, Sleep Apnea, and Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Gerald M Reaven, Professor Emeritus, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 5U01HL108647-04 (NIH)
Record Dates: First submitted 2014-07-07; First posted 2014-07-17 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Insulin Sensitivity; Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; insulin sensitivity; cardiovascular risk; positive airway pressure therapy
MeSH Terms: conditions — Insulin Resistance; Sleep Apnea, Obstructive | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pioglitazone (Active Comparator): pioglitazone 45 mg, oral, daily
  Interventions: Drug: Pioglitazone
- placebo (Placebo Comparator): Placebo, one pill daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Pioglitazone — 45 mg daily Insulin sensitizing
  Other Names: actos
  Arms: pioglitazone
Drug: placebo — Compare with pioglitazone
  Arms: placebo

SUMMARY:
Obstructive sleep apnea (OSA) and type 2 diabetes confer increasing economic, social, and public health burdens in the United States. That these diseases appear to co-exist and together increase one's risk of cardiovascular disease renders investigation into their shared pathophysiology even more urgent. Investigators will assess prevalence of insulin resistance, a precursor to diabetes, among overweight patients with OSA. Among those at highest risk of diabetes, investigators will randomize participants to pioglitazone or placebo to see the efficacy of the intervention on improving OSA, insulin resistance, and/or insulin secretion. In a separate intervention, investigators will evaluate the cardiometabolic benefits of continuous positive airway pressure (CPAP) for 12 weeks in patients with OSA. Investigators will also study subjects from the community without known sleep apnea, and assess whether insulin-resistant individuals are at risk for sleep apnea using clinical screening questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Individuals
* Age 30-70 years old
* BMI- 25-40 kg/m2
* Must meet criteria for obstructive sleep apnea by overnight in-laboratory polysomnography

Exclusion Criteria:

* Any significant co-morbidities, such as diabetes, active heart, kidney, liver diseases, or active or history of bladder cancer.
* Must not have previously received treatment for OSA, including CPAP.
* Must not be receiving any medications intended for weight loss, or those known to influence insulin sensitivity.
* Pregnancy/lactation is also an exclusion.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-09; Primary Completion 2014-07 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald M Reaven, M.D., Principal Investigator — Stanford University

REFERENCES:
- [Derived] Liu A, Kim SH, Ariel D, Abbasi F, Lamendola C, Cardell J, Xu S, Patel S, Tomasso V, Mojaddidi H, Grove K, Tsao PS, Kushida CA, Reaven GM. Does enhanced insulin sensitivity improve sleep measures in patients with obstructive sleep apnea: a randomized, placebo-controlled pilot study. Sleep Med. 2016 Jun;22:57-60. doi: 10.1016/j.sleep.2016.06.005. Epub 2016 Jun 21. PMID 27544837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Dates: July 10 2010 - March 2014
Period: Overall Study
Arm/Group | Pioglitazone | Placebo
Started | 30 | 15
Completed | 30 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Placebo | Total
Number analyzed (Participants) | 30 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (11) | 50 (12) | 50.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 20 | 10 | 30
Changes in sleep measure [Mean (Standard Deviation); unit: Apnea-hypopnea index (AHI) events/hour] — apnea-hypopnea index (AHI) events per hour
  Apnea-hypopnea index (AHI) events/hour | 36.9 (11.9) | 40.8 (12.3) | 38.9 (12.1)
Insulin Sensitivity [Mean (Standard Deviation); unit: mmol/L] — Steady-state plasma glucose (mmol/L)
  mmol/L | 11.9 (2.1) | 12.3 (2.0) | 12.1 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Apnea-hypopnea Index (AHI) Outcome Measure in Response to Pioglitazone or Placebo
Description: To evaluate the effects of pioglitazone versus placebo on AHI in patients with OSA.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: AHI events/hour
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 30 | 15
AHI events/hour | 35.8 [21 to 49] | 34.4 [18 to 47]

ADVERSE EVENTS:
Arm/Group | Pioglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/15
Other Adverse Events (participants affected / at risk) | 2/30 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=30) | Placebo (N=15)
weight gain (Product Issues) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Unrecognized adverse effect of pioglitazone could have obviated a beneficial effect of enhanced insulin sensitivity on OSA related sleep measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes